CLINICAL TRIAL: NCT01085006
Title: The Effect of Tranexamic Acid Administration on Postpartum Hemorrhage During and After Cesarean Delivery
Brief Title: The Effect of Tranexamic Acid on Postpartum Hemorrhage During and After Cesarean Delivery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Laleh Eslamian/ Associated professor/obstetrician &gynecologist, Associated Prof
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 830
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-11

CONDITIONS: Hemorrhage
Keywords: cesarean delivery; Tranexamic acid; hemorrhage; Spinal analgesia; 1-the amount of hemorrhage during cesarean delivery; 2-the amount of hemorrhage in the first 2 hours of cesarean delivery; 3-the amount of hemorrhage in the first 24 hour after cesarean delivery
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Experimental)
  Interventions: Drug: Tranexamic acid
- normal saline infusion (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic acid in cases, normal saline in controls
  Arms: Tranexamic acid
Drug: Normal saline — Tranexamic acid in cases, normal saline in controls
  Arms: normal saline infusion

SUMMARY:
Intravenous Tranexamic acid is used to reduce the hemorrhage during and after cesarean delivery in a double blind randomized placebo controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Term pregnancy
2. Single fetus
3. Maximally only one previous cesarean delivery

Exclusion Criteria:

1. More than one previous cesarean delivery
2. Hx of other abdominal or pelvic surgery
3. Hx of medical disorders
4. Hx of thromboembolic disorders
5. Polyhydramnios
6. Macrosomia
7. Preeclampsia
8. Hx of sensitivity to Tranexamic acid
9. Abnormal Pt, PTT, PT or INR

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laleh Eslamian, MD, Principal Investigator — Associated Prof, Obstetrician & Gynecologist
Locations (1):
- Laleh Eslamian, Tehran, Iran

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid | Normal Saline Infusion
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Normal Saline Infusion | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27 (3.4) | 27.6 (4.1) | 27.3 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: The Amount of Hemorrhage During Cesarean Delivery and Within 2 Hours Afterward
Time Frame: During the procedure and within 2 hours afterwards
Measure: Median (Full Range); unit: ml
Arm/Group | Tranexamic Acid | Normal Saline Infusion
Number analyzed (Participants) | 50 | 50
ml | 260 [200 to 350] | 380 [200 to 560]

2. Secondary Outcome: Amount of Hemorrhage in the First 24 Hour After Cesarean Delivery
Time Frame: First 24 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Tranexamic Acid | Normal Saline Infusion
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes